CLINICAL TRIAL: NCT06284486
Title: A Multi-Site Break Through Cancer Trial: Phase II Study Investigating Dual Inhibition of BCL2 and Menin in AML MRD Using the Combination of Venetoclax and Revumenib
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Syndax Pharmaceuticals (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0794; NCI-2024-01721 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; revumenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax + Revumenib (Experimental): Participants may receive the combination of venetoclax and revumenib for up to 1 year, and then 1 more year of venetoclax alone. You will no longer be able to take the study drug(s) if the disease gets worse or if intolerable side effects occur. Participants will take venetoclax by mouth on 1 time a day at about the same time each day, on Days 1-14 of each cycle. Take each dose with about 1 cup of water within 30 minutes after a meal, preferably breakfast.
  Interventions: Drug: Venetoclax; Drug: Revumenib

INTERVENTIONS:
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Revumenib — Given by PO
  Other Names: SNDX-5613

SUMMARY:
To learn if the combination of venetoclax and revumenib can help to control MRD-positive AML.

DETAILED DESCRIPTION:
Primary Objectives

* Phase I: To determine the safety, tolerability, and recommended phase II dose (RP2D) of the combination of revumenib and venetoclax for patients with acute myeloid leukemia (AML) and detectable minimal or measurable residual disease (MRD).
* Phase II: To assess the efficacy of the combination of venetoclax and revumenib in clearance of MRD in patients with AML.

Secondary Objectives

* To assess overall survival (OS), relapse-free survival (RFS), event-free survival (EFS) and duration of response (DOR).
* To determine clinical flow and genetic MRD concordance rate

Exploratory Objectives

* To evaluate molecular and cellular markers that may be predictive of antitumor activity and/or resistance.
* To correlate MRD negativity with clinical outcomes (survival and relapse risk)
* To evaluate concordance of standard and novel MRD assays
* To explore the safety and activity of venetoclax plus revumenib in the pediatric population

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years with weight ≥ 45Kg.
2. ECOG performance status of ≤ 2. (if aged ≥18 years); Karnofsky Performance Scale of ≥50 (if aged ≥16 years and <18 years); Lansky Performance Score of ≥50 (if aged <16 years).
3. Leukemia status:

   * Known history of NPM1mt, or KMT2Ar, or NUP98r AML.
   * Bone marrow assessment showing no leukemia by morphology (blasts <5%) in first remission following high intensity chemotherapy or at least 2 cycles of low intensity therapy (e.g. hypomethylating agent or low-dose cytarabine-based), or in second remission following any therapy, with MRD ≥ 0.1% identified by multiparameter flow cytometry using central lab testing.
   * No clinically active extramedullary disease.
4. Baseline ejection fraction must be > 40%.
5. Adequate hepatic function (direct bilirubin < 1.5x upper limit of normal (ULN) unless increase is due leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
6. Adequate renal function with an estimated glomerular filtration rate ≥ 60 mL/min based on local institutional practice for age-appropriate determination.
7. Able to swallow pills.
8. Participants or parent/guardian is willing and able to provide informed consent. Interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy, whichever is shorter. Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
9. Women of childbearing potential must agree to adequate methods of contraception during the study and at least 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study and at least 3 months after the last treatment.

Exclusion Criteria:

1. Prior treatment with a menin inhibitor.
2. Participants who are expected to receive standard therapy (either intensive or hypomethylating agent and venetoclax) with continued tolerability and benefit.
3. Participants who are expected to be able to proceed with stem cell transplantation within the next 30 days.
4. Participants with any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the patient at unacceptable risk of study treatment.
5. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for patients with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
6. Participants with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
7. Participants with a concurrent active malignancy under treatment.
8. Known active hepatitis B (HBV) or Hepatitis C (HCV) or HIV infection.
9. Female subjects who are pregnant or breast-feeding.
10. Participant has an active uncontrolled infection.
11. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
12. QTc >450 msec for males and QTc >470 msec for females using the Fridericia Formula.
13. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the participants's participation for the full duration of the study, or is not in the best interest of the patient to participate.
14. Clinically active central nervous system (CNS) leukemia.
15. Participants on immunosuppressive therapy post-HSCT at the time of screening (must be off all systemic immunosuppression therapy for at least 2 weeks and calcineurin inhibitors for at least 4 weeks). The use of topical steroids for cutaneous graft-versus-host disease (GVHD) or stable systemic steroid doses less than or equal to 20 mg of prednisone daily are permitted.
16. Participants with Grade > 2 active acute GVHD, moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ghayas Issa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org